CLINICAL TRIAL: NCT01348399
Title: Evaluation of Effectiveness and Safety of XIENCE PRIME™ in Routine Clinical Practice; A Multicenter, Prospective Observational Study
Brief Title: Evaluation of Effectiveness and Safety of XIENCE PRIME Stent (IRIS-PRIME)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2011-01
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease requiring drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- XIENCE PRIME stents

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of XIENCE PRIME stent in the "real world" daily practice as compared with other drug eluting stents (DESs)

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, open-label registry to compare the effectiveness and safety of XIENCE PRIME stents versus other DESs in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving XIENCE PRIME stents.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients presented with cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving XIENCE PRIME stents.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or target- Vessel Revascularization (TVR) | 12 months post procedure

SECONDARY OUTCOMES:
Death (all cause and cardiac) | one month
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | yearly up to 5 years
MI | one month
MI | 6 months
MI | yearly up to 5 years
Composite of death or MI | one month
Composite of death or MI | 6 months
Composite of death or MI | yearly up to 5 years
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | yearly up to 5 years
TVR | one month
TVR | 6 months
TVR | yearly up to 5 years
Target-lesion revascularization (TLR) | one month
Target-lesion revascularization (TLR) | 6 months
Target-lesion revascularization (TLR) | yearly up to 5 years
Stent thrombosis (ARC criteria) | one month
Stent thrombosis (ARC criteria) | 6 months
Stent thrombosis (ARC criteria) | yearly up to 5 years
Procedural success (defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization) | At discharge from the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center; Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea
Locations (29):
- South Korea (29):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang Univ. Bucheon Hospital, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Presbyterian Medical Center, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Kwangju Christian Hospital, Kwangju
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Bundang Cha Medical Center, Seongnam
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan